CLINICAL TRIAL: NCT01897012
Title: A Phase 1 Trial of MLN8237 Plus Romidepsin for Relapsed/Refractory Aggressive B-Cell and T-Cell Lymphomas
Brief Title: Alisertib and Romidepsin in Treating Patients With Relapsed or Refractory B-Cell or T-Cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01272; NCI-2013-01272 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); TX035; 2012-0602; 9342 (Other: M D Anderson Cancer Center); 9342 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH); UM1CA186688 (NIH)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: MYC Positive; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Burkitt Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Mature T- and NK-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Burkitt Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory Hodgkin Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Hodgkin Disease; Lymphoma, Mantle-Cell; Lymphoma, T-Cell | interventions — MLN 8237; romidepsin; Depsipeptides; Lactones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (alisertib, romidepsin) (Experimental): Patients receive alisertib PO BID on days 1-7 (dose levels 1-4) or days 1-3, 8-10, and 15-17 (dose levels 5-8). Patients also receive romidepsin IV over 4 hours on days 1 and 8 (dose levels 1-4) or 2, 9, and 16 (dose levels 5-8). Treatment repeats every 21 days (dose levels 1-4) or 28 days (dose levels 5-8) for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis; Drug: Romidepsin

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Romidepsin — Given IV
  Other Names: Antibiotic FR 901228; Depsipeptide; FK228; FR901228; Istodax; N-[(3S,4E)-3-Hydroxy-7-mercapto-1-oxo-4-heptenyl]-D-valyl-D-cysteinyl-(2Z)-2-amino-2-butenoyl-L-valine, (4->1) Lactone, Cyclic

SUMMARY:
This phase I trial studies the side effects and best dose of alisertib and romidepsin in treating patients with B-cell or T-cell lymphomas that have returned after a period of improvement (relapsed) or have not responded to treatment (refractory). Alisertib and romidepsin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety profile of alisertib (MLN8237) plus romidepsin. II. To determine the maximum tolerated dose (MTD), if reached, of MLN8237 administered in combination with romidepsin.

SECONDARY OBJECTIVES:

I. To evaluate objective response rate (ORR) and complete response (CR) of the combined regimen.

II. To assess whether higher levels of expression of aurora kinase A correlate with outcomes.

III. To determine if this combination results in downregulation of targets of v-myc myelocytomatosis viral oncogene homolog (avian) (C-Myc) in C-Myc positive patients, induces mitotic catastrophe, changes immune system or other host responses, or upregulates markers for apoptosis.

OUTLINE: This is a dose-escalation study.

Patients receive alisertib orally (PO) twice daily (BID) on days 1-7 (dose levels 1-4) or days 1-3, 8-10, and 15-17 (dose levels 5-8). Patients also receive romidepsin intravenously (IV) over 4 hours on days 1 and 8 (dose levels 1-4) or 2, 9, and 16 (dose levels 5-8). Treatment repeats every 21 days (dose levels 1-4) or 28 days (dose levels 5-8) for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed Hodgkin lymphoma, Burkitt's lymphoma, double-hit lymphoma, other c-Myc positive B-cell lymphoma, diffuse large-B cell lymphoma including those patients with history of transformed follicular lymphoma, mantle cell lymphoma, or peripheral T-cell lymphoma
* Patients must have at least one 1.5 cm bidimensional measurable lesion
* Relapsed or refractory after at least 1 front-line therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Direct bilirubin =< 1 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< 2 x institutional upper limits of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of MLN8237 plus romidepsin administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MLN8237 plus romidepsin administration
* Ability to understand and the willingness to sign a written informed consent document
* According to current guidelines, patients must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration; these guidelines may change pending results from an ongoing food effects study

Exclusion Criteria:

* Patients who have had chemotherapy, radiation therapy, or other investigational agents within 3 weeks prior to entering study, 6 weeks for nitrosoureas or mitomycin
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN8237, including but not limited to established allergic reaction to benzodiazepines, or romidepsin; agents that alter gastric pH may change MLN8237 absorption are not permitted; proton pump inhibitors need to be stopped 4 days prior to the first dose of MLN8237; histamine-2 (H2) receptor antagonists are not permitted from the day prior (day -1) through to the end of MLN8237 dosing; antacid preparations are not permitted for 2 hours before or 2 hours after administration of MLN8237
* Co-administration of enzyme-inducing antiepileptic drugs, rifampin, rifabutin, rifapentine, or St. John's wort is not permitted; concurrent bisphosphonate therapy is allowed if it was started before study entry and is maintained at recommended dosing intervals; bisphosphonate therapy may not be initiated after study entry
* Any serious active disease or co-morbid condition, which in the opinion of the principal investigator, will interfere with the safety or compliance of the trial
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MLN8237 and/or romidepsin
* Ejection fraction (EF) < 40% or myocardial infarction (MI) within the past 3 months; known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen; or any conditions that could result in excessive toxicity associated with the benzodiazepine-like effects of MLN8237
* Requirement for constant administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes; intermittent uses of antacids or H2 antagonists are allowed
* Inability to swallow oral medication or to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration or any condition that would modify small bowel absorption of oral medications, including malabsorption, or resection of pancreas or upper bowel; treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine, oxcarbazepine, primidone or phenobarbital, or rifampin, rifabutin, rifapentine, or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study; patients must be cautiously co-medicated with agents that cause corrected QT interval (QTc) prolongation and agents that are strong or moderate enzyme inhibitors during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (utilized for adverse event reporting beginning April 1, 2018) | Up to 4 weeks post-treatment
Maximum tolerated dose graded according to NCI CTCAE version 5.0 | Up to 28 days
  Maximum tolerated dose is defined as the highest dose level at which 6 patients have been treated with fewer than 2 instances of dose-limiting toxicities.

SECONDARY OUTCOMES:
Overall response rate | Up to 4 weeks post-treatment
  Point estimates along with 95% confidence intervals will be provided.
Complete response | Up to 4 weeks post-treatment
  Point estimates along with 95% confidence intervals will be provided.

OTHER OUTCOMES:
Aurora A kinase expression intensity, assessed by immunohistochemistry | Baseline
  Will be correlated with response.
Change in gene expression profiles | Baseline to up to 28 days (course 1)
  Will be correlated with response.

CONTACTS AND LOCATIONS:
Overall Officials: Hun Lee, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States